CLINICAL TRIAL: NCT04038827
Title: Search of Circulating Endothelial Cells of Donor Origin After Allogeneic Hematopoietic Stem Cell Transplantation: Evaluation for Potential Clinically Relevant Implications in the Context of Graft-Versus-Host Disease
Brief Title: Origin of CEC in Patients After Allo-HSCT
Acronym: DCEC-PIANO
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Università degli Studi di Brescia (Other); University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Camillo Almici MD, Director of the Stem Cells Lab, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: 0037975
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Graft Versus Host Disease, Acute; Endothelial Dysfunction; Immune Tolerance
Keywords: Circulating Endothelial Cells; Graft versus Host Disease; Neovascularization; Allotransplantation
MeSH Terms: conditions — Graft vs Host Disease; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be obtained from each single CEC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: D-CEC counting — By means of preliminary bulk separation step with the CellSearch system, single CEC will be sorted

SUMMARY:
We believe that CEC, besides coming from cells shedding from patient vasculature, could partly belong to donor, originating from the cellular graft.

DETAILED DESCRIPTION:
In consideration of the fact that the vascular endothelium has been shown to be a target of GvHD in early stage and that the count of CEC represent a marker of endothelial damage, we want to correlate the presence of donor CEC at engraftment with a putative protective function against GVHD manifestations. We will enroll patients affected by hematologic disorders undergoing allo-HSCT. At time of engraftment and at + 3 months after allo-HSCT, CEC identified and counted by means of the CellSearch system, will be recovered from the counting cartridge and further sorted at the single cell level. STR profile of each single CEC recovered will be performed in order to define host versus donor origin of each CEC analysed.

Through the conduct of this study, we expect to upfront identify patients who will or will not manifest GvHD. This result will allow definitely different clinical approaches: stringent monitoring and early therapeutic intervention, before refractory disease's development, in the formers, while, sparing unnecessarily expensive testing or heavier treatment in the latters.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing allo-HSCT for their neoplastic hematologic diseases
* written informed consent
* achievement of hematopoietic recovery from aplasia post-allo-HSCT
* predictable life expectancy > 6 months

Exclusion Criteria:

* presence of active malignant hematologic disease at time of allo-HSCT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing allo-HSCT for their neoplastic hematologic disorders
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Presence of D-CEC at time of engraftment in patients undergoing allo-HSCT | Within 30 days from allo-HSCT
  Single CEC will be isolated and STR profile determined
Correlate presence/absence of D-CEC with GVHD manifestations | day +100 post allo-HSCT
  D-CEC presence will be correlated with GVHD onset

SECONDARY OUTCOMES:
Presence of donor CEC embedded in the endothelial layer of patients microvasculature at late timepoint after allo-HSCT | day +100 post allo-HSCT
  CISH analysis will be performed on tissue biopsies at 3 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Almici, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analyzed during the current study will be available from the corresponding author on reasonable request after publication of results
Supporting Information: Study Protocol, ICF
Time Frame: after publication of results
Access Criteria: Request to Principal Investigator

REFERENCES:
- [Background] Penack O, Socie G, van den Brink MR. The importance of neovascularization and its inhibition for allogeneic hematopoietic stem cell transplantation. Blood. 2011 Apr 21;117(16):4181-9. doi: 10.1182/blood-2010-10-312934. Epub 2011 Jan 21. PMID 21258010
- [Background] Riesner K, Shi Y, Jacobi A, Krater M, Kalupa M, McGearey A, Mertlitz S, Cordes S, Schrezenmeier JF, Mengwasser J, Westphal S, Perez-Hernandez D, Schmitt C, Dittmar G, Guck J, Penack O. Initiation of acute graft-versus-host disease by angiogenesis. Blood. 2017 Apr 6;129(14):2021-2032. doi: 10.1182/blood-2016-08-736314. Epub 2017 Jan 17. PMID 28096092
- [Background] Fadini GP, Avogaro A. Cell-based methods for ex vivo evaluation of human endothelial biology. Cardiovasc Res. 2010 Jul 1;87(1):12-21. doi: 10.1093/cvr/cvq119. Epub 2010 Apr 28. PMID 20427336
- [Background] Lanuti P, Rotta G, Almici C, Avvisati G, Budillon A, Doretto P, Malara N, Marini M, Neva A, Simeone P, Di Gennaro E, Leone A, Falda A, Tozzoli R, Gregorj C, Di Cerbo M, Trunzo V, Mollace V, Marchisio M, Miscia S. Endothelial progenitor cells, defined by the simultaneous surface expression of VEGFR2 and CD133, are not detectable in healthy peripheral and cord blood. Cytometry A. 2016 Mar;89(3):259-70. doi: 10.1002/cyto.a.22730. Epub 2015 Aug 25. PMID 26305912
- [Background] Lanuti P, Simeone P, Rotta G, Almici C, Avvisati G, Azzaro R, Bologna G, Budillon A, Di Cerbo M, Di Gennaro E, Di Martino ML, Diodato A, Doretto P, Ercolino E, Falda A, Gregorj C, Leone A, Losa F, Malara N, Marini M, Mastroroberto P, Mollace V, Morelli M, Muggianu E, Musolino G, Neva A, Pierdomenico L, Pinna S, Piovani G, Roca MS, Russo D, Scotti L, Tirindelli MC, Trunzo V, Venturella R, Vitagliano C, Zullo F, Marchisio M, Miscia S. A standardized flow cytometry network study for the assessment of circulating endothelial cell physiological ranges. Sci Rep. 2018 Apr 11;8(1):5823. doi: 10.1038/s41598-018-24234-0. PMID 29643468
- [Background] Almici C, Skert C, Verardi R, Di Palma A, Bianchetti A, Neva A, Braga S, Malagola M, Turra A, Marini M, Russo D. Changes in circulating endothelial cells count could become a valuable tool in the diagnostic definition of acute graft-versus-host disease. Transplantation. 2014 Oct 15;98(7):706-12. doi: 10.1097/TP.0000000000000385. PMID 25119132
- [Background] Almici C, Skert C, Bruno B, Bianchetti A, Verardi R, Di Palma A, Neva A, Braga S, Piccinelli G, Piovani G, Malagola M, Bernardi S, Giaccone L, Brunello L, Festuccia M, Baeten K, Russo D, Marini M. Circulating endothelial cell count: a reliable marker of endothelial damage in patients undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2017 Dec;52(12):1637-1642. doi: 10.1038/bmt.2017.194. Epub 2017 Sep 11. PMID 28892085
- [Background] Almici C, Neva A, Skert C, Bruno B, Verardi R, Di Palma A, Bianchetti A, Braga S, Piovani G, Cancelli V, Omede P, Baeten K, Rotta G, Russo D, Marini M. Counting circulating endothelial cells in allo-HSCT: an ad hoc designed polychromatic flowcytometry-based panel versus the CellSearch System. Sci Rep. 2019 Jan 14;9(1):87. doi: 10.1038/s41598-018-36442-9. PMID 30643152
- [Background] Cortesini R, Suciu-Foca N. ILT3+ ILT4+ tolerogenic endothelial cells in transplantation. Transplantation. 2006 Jul 15;82(1 Suppl):S30-2. doi: 10.1097/01.tp.0000231437.12890.64. PMID 16829792
- [Background] Taflin C, Charron D, Glotz D, Mooney N. Regulation of the CD4+ T cell allo-immune response by endothelial cells. Hum Immunol. 2012 Dec;73(12):1269-74. doi: 10.1016/j.humimm.2012.07.009. Epub 2012 Jul 16. PMID 22813652
- [Background] Pober JS. Is host endothelium a silver lining for allografts? Lancet. 2001 Jan 6;357(9249):2-3. doi: 10.1016/S0140-6736(00)03558-3. No abstract available. PMID 11197355
- [Background] Wu SR, Reddy P. Tissue tolerance: a distinct concept to control acute GVHD severity. Blood. 2017 Mar 30;129(13):1747-1752. doi: 10.1182/blood-2016-09-740431. Epub 2017 Feb 2. PMID 28153825
- [Background] Lin Y, Weisdorf DJ, Solovey A, Hebbel RP. Origins of circulating endothelial cells and endothelial outgrowth from blood. J Clin Invest. 2000 Jan;105(1):71-7. doi: 10.1172/JCI8071. PMID 10619863